CLINICAL TRIAL: NCT00650026
Title: Multicenter Early Access Program of the Safety of Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Active Rheumatoid Arthritis
Brief Title: Early Access Program of the Safety of Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Active Rheumatoid Arthritis
Acronym: ReAct
Status: Approved for marketing | Type: Expanded Access
Sponsor: Abbott (Industry)
Responsible Party: Larry McNamee, Sr. Clinical Research Manager, Abbott
Other Study IDs: M03-583
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

INTERVENTIONS:
Biological: adalimumab — 40 mg adalimumab every other week
  Other Names: ABT-D2E7; Humira

SUMMARY:
Multicenter Early Access Program of the Safety of Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects with Active Rheumatoid Arthritis

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years or older
* Females - post-menopausal for at least 1 year, surgically sterile or practicing an acceptable method of birth control
* Females - negative pregnancy test at screening
* Confirmed diagnosis of active RA >= 6 swollen joints and >= 9 tender joints
* Met ACR criteria for diagnosis of RA for at least 3 months
* Active RA defined by a DAS >= 3.2 at study entry

Exclusion Criteria:

* Subject had prior treatment with cyclophosphamide or chlorambucil
* Subjects previously treated with total lymphoid irradiation or anti-CD4 or CAMPATH 1H monoclonal antibodies resulting in CD4 lymphopenia
* Prior treatment with intravenous immunoglobulin or investigational agent in with 30 days or 5 half-lives of adalimumab
* Subject with history of cancer within the past 10 years other than resected basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult